CLINICAL TRIAL: NCT00772408
Title: Relationship Between TLR2 Polymorphism and Pulmonary Tuberculosis
Brief Title: Toll-like Receptor 2 Gene Polymorphism, Serum Cytokines and Susceptibility to Disease Severity or Treatment Response of Pulmonary Tuberculosis
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NSC 95-2314-B-182A-030
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2008-10

CONDITIONS: Pulmonary Tuberculosis; Genetic Variants of Host; Immune Response of Host
Keywords: pulmonary tuberculosis; Toll-like receptor 2 gene polymorphisms; blood lymphocyte subsets; systemic symptoms; pleural effusion
MeSH Terms: conditions — Tuberculosis, Pulmonary; Pleural Effusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood leukocyte DNA and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TB: patients with pulmonary TB
- control: healthy controls

SUMMARY:
Infection with Mycobacterium tuberculosis remains at epidemic levels globally. Innate and adaptive immune responses evolve as protective mechanisms against mycobacterial infection in humans. Toll-like receptors (TLRs) are transmembrane proteins characterized by an extracellular leucine-rich domain that participates in ligand recognition and an intracellular tail. TLRs are the first defense system to detect potential pathogens, initiate immune responses and form the crucial link between innate and adaptive immune systems. Stimulation of TLR initiates a signaling cascade that involves a number of proteins, such as MyD88 and IL-1 receptor-associated kinase. This signal cascade leads to NF-κB activation, which induce the secretion of pro-inflammatory cytokines.

TLR2 is a family of TLR family and has been reported to be the principle mediator of macrophage activation in response to mycobacterium. Growing amounts of data suggest that the ability of certain individuals to respond properly to TLR ligands may be impaired by single nucleotide polymorphisms (SNPs) within TLR genes, resulting in an altered susceptibility to, or course of, infectious disease. The genetic polymorphism of TLR2 (arginine to glutamine substitution at residue 753 (Arg753Gln)) has been associated with a negative influence on TLR2 function, which may, in turn, determine the innate host response to mycobacteria. In addition, another polymorphism (Arg677Trp) of the TLR2 was reported to be associated with susceptibility to tuberculosis in Tunisian patients. Moreover, in Mycobacterium leprosy patients with TLR2 mutation (Arg677Trp), production of IL-2, IL-12, IFN-gamma, and TNF-alpha by M. leprae-stimulated peripheral blood mononuclear cell were decreased compared with that in groups with wild-type TLR2.

To date, there have been no studies of the association of SNPs of TLR2 with cytokine profiles and clinical outcomes on M. tuberculosis. We hypothesize that polymorphisms in the TLR2 are associated with :

1. increased prevalence of active pulmonary TB infection,
2. altered levels of pro-inflammatory and anti-inflammatory cytokines in serum,
3. clinical outcomes and presentations. We thus design a prospective case-control study to test this hypothesis. The frequency of TLR2 polymorphisms in both pulmonary TB patients and healthy controls will be determined by polymerase chain reaction-restriction fragment length polymorphism. Serial serum levels of IL-12, IFN-γ, and IL-10 in pulmonary TB patients with or without TLR2 polymorphisms will be measured by enzyme linked immunosorbent assay. Relationships between TLR2 polymorphisms and serum cytokines dynamics or clinical outcomes will be analyzed.

DETAILED DESCRIPTION:
Infection with Mycobacterium tuberculosis (TB) remains at epidemic levels globally. One third of the word's population is infected with this organism, making tuberculosis the most prevalent infectious disease. Annually, 8 million people contract the disease, and there are 2 million deaths worldwide each year, with increasing prevalence predicted over the next several decades.(1) In Taiwan, there are 24,161 reporting cases registered in the national tuberculosis database, and 17,660 were diagnosed as confirmed TB cases in 2004. The annual incidence rate of newly TB cases is 74.11 per 100,000 people.

Immunity Against Mycobacteria M. tuberculosis is a unique pathogen in that once infection occurs, even in the face of in intact host immune system it is not eradicated but establishes a chronically persistent, or latent, state. Viable organisms remain sequestered by the host's immune system, though they fail to progressively replicate. Subsequently, in approximately 15 % of those latently infected, the infection may reactivate with the development of overt, progressive, pulmonary disease. Impairments in the immune system may linked to reactivation, but much remains to be discovered about control of infection by M. tuberculosis.

Innate and adaptive immune responses evolve as protective mechanisms against infectious organisms in humans. Phagocytosis of relatively small numbers of organisms initiated the host response in the alveolar cells.CD14 and toll-like receptors (TLRs) are examples of pattern recognition receptors that detect antigenic molecules on the surface of bacteria and mycobacteria.(2) The family of TLRs is capable of recognizing conserved microbial patterns including components of bacterial cell wall, microbial nucleic acids, and bacterial motility. TLRs are the first defense system to detect potential pathogens, initiate immune responses and form the crucial link between innate and adaptive immune systems. TLRs also play an import role in the pathophysiology of infectious diseases, inflammatory diseases such as Crohn's disease and atherosclerosis, possibly play a role in autoimmune disease.( 3) TLRs are transmembrane proteins characterized by an extracellular leucine-rich domain that participates in ligand recognition and an intracellular tail that contains a conserved region called the Toll interleukin 1 receptor (IL-1R) homology domain.(4) Stimulation of TLR initiates a signaling cascade that involves a number of proteins, such as MyD88 and IL-1 receptor-associated kinase.(5) This signal cascade leads to NF-κB activation, which induce the secretion of pro-inflammatory cytokines. TLR2 has been reported to be the principle mediator of macrophage activation in response to mycobacteria. TLR2 expression is found primarily on alveolar macrophages and epithelial cells type Ⅱwithin tuberculous granulomas. Due to its ability to recognize Mycobacterium tuberculosis and its components, the expression of TLR2 at the site of disease is critical. (6, 7)

Single nucleotide polymorphisms of Toll-like receptors and susceptibility to pulmonary tuberculosis Growing amounts of data suggest that the ability of certain individuals to respond properly to TLR ligands may be impaired by single nucleotide polymorphisms (SNPs) within TLR genes, resulting in an altered susceptibility to, or course of, infectious disease.TLR2 is a member of the TLR family.(8) Animal studies have shown that TLR2-knockout mice are more susceptible to septicemia due to Staphylococcus and Listeria monocytogenes, meningitis due to Streptococcus pneumoniae, and infection with Mycobacterium tuberculosis, suggesting the functional TLR2 polymorphisms may impair host response to a certain spectrum of microbial pathogens.(9) Mycobacterium tuberculosis infects 2 billion people globally, yet only 10 % develop clinical disease. The identification of factors that predispose to disease could aid the development of new therapies and vaccines.

The genetic polymorphism of TLR2 (arginine to glutamine substitution at residue 753 (Arg753Gln)) has been associated with a negative influence on TLR2 function, which may, in turn, determine the innate host response to mycobacteria. In a recent cohort study, this polymorphism was demonstrated to influence the risk of developing tuberculosis in Turkey patients.(10) In addition, another polymorphism (Arg677Trp) of the TLR2 was reported to be associated with susceptibility to tuberculosis in Tunisian patients (11), as well as lepromatous leprosy(12). More recently, polymorphisms in CD 14 and TLR2 are demonstrated to be associated with increased prevalence of infection in critical ill adults (13). TLR2 gene Arg753Lin polymorphism is also strongly associated with rheumatic fever in children. Moreover, this polymorphism is a risk factor for coronary restenosis.(14)

Dynamics of cytokine generation by inflammatory cells and clinical outcomes TLRs mediate the activation of cells of the innate immune system leading to dynamic functions including direct anti-microbial activity, induction of cytokine secretion, triggering dendritic cell maturation, and triggering apoptosis. Macrophage phagocytosis of M. tuberculosis is accompanied by activation of the transcription factor NF-κB and secretion of inflammatory mediators that play an important role in granuloma formation and immune protection. Once antigen-presenting cells (alveolar macrophage or dendritic cell) have processed the engulfed mycobacterial protein, they present the antigens in the context of major histocompatibility complex (MHC) class Ⅱ surface molecules to naïve CD4+ lymphocytes. The antigen-presenting cell produce IL-12 to bias the immune reaction to T helper 1 (Th1) and IL-1, which stimulate the CD4+ lymphocytes to produce IL-2. The net result is the rapid clonal expansion of specific CD4+ Th1 lymphocyte, which produce interferon gamma (IFNγ), a cytokine that activate the macrophage that have engulfed mycobacteria to become mycobactericidal. It has been demonstrated that a 19-kDa lipoprotein of M.tb triggered cells to activate NF-κB and secret IL-2 in a TLR-2 dependent pathway(15).On the other hand, The Th2 cytokines may play roles in mycobacterial inflammation as well. IL-10, produced by monocytes, macrophage, and lymphocytes, is upregulated after mycobacterail infection, and downregulates IFN-γ production. Secretion of IL-10 will favor the activation of a Th2 response which is incapable of destroying intracellular pathogens. Activation of human monocyte derived dendritic cells with M.tb 19 kDa lipoprotein results in the preferential secretion of IL-12 over IL-10 (16, 17).

The balance between IFN-γ and IL-10 production may determine wheather effective immunity is established or anergy supervenes in any infected patient, and may influence clinical outcome. Levels of IFN-γ are higher in moderate disease than advanced diaseses, whereas advanced cases showed higher IL-12, and TNF-alpha compared with cases of moderate TB. In most patients, decreased interferon-γ production by PBMC seems to be a transient response because it is significantly increased in most active TB patients during and following successful therapy. In the TB patients with a systemic reaction, both IL-12 and IFN-γproduction by monocytes after challenge with a virulent M.tb strain were significantly reduced compared to PPD reactor group. Bronchoalveolar lavarge fluid levels of IFN-γ was also correlated with disease grading and decreased after anti-TB chemotherapy(18).However, some patients remain anergic in vivo and in vitro after chemotherapy, and the underlying biochemical mechanisms for T cell anergy in modulating protection or pathology in TB needs further clarification.(19)

Toll-like receptor 2 mutation and the profiles of cytokines The production of IL-6 and IL-10 from dendritic cells in response to M.tuberculosis is principally dependent on TLR2 (20). On the other hand, M. tuberculosis can induce IL-12 production in the absence of either TLR2 or TLR4. In leprosy patients with TLR2 mutation (Arg677Trp), production of IL-2, IL-12, IFN-gamma, and TNF-alpha by M. leprae-stimulated peripheral blood mononuclear cell were decreased compared with that in groups with wild-type TLR2. However the cells from patients with the TLR2 mutation showed significantly increased production of IL-10. These results suggest that TLR2 signal pathway plays a critical role in the alteration of cytokine profiles in PBMC from patients with mycobacterial infection. ( 21)

In summary, TLR2 polymorphisms have been shown to be associated with susceptibility to tuberculosis in Turkey and Tunisian people. These polymorphisms have been demonstrated to affect cytokine production by monocytes in vitro. To date, there have been no studies of the association of SNPs of TLR2 with serum cytokine profiles and clinical outcomes on M. tuberculosis infection. We hypothesize that polymorphisms in the TLR2 are associated with :

1. increased prevalence of active pulmonary TB infection,
2. altered levels of pro-inflammatory and anti-inflammatory cytokines in serum,
3. clinical outcomes and presentations. We thus design a prospective case control study to test this hypothesis. The frequency of TLR2 polymorphisms in both pulmonary TB patients and healthy controls will be determined and compared by polymerase chain reaction-restriction fragment length polymorphism. Serial serum levels of IL-12, IFN-γ, and IL-10 in pulmonary TB patients with or without TLR2 polymorphisms will be measured by enzyme linked immunosorbent assay at initial presentation, 2months and 6 months after anti-TB drugs treatment. Relationships between TLR2 polymorphisms and serum cytokines dynamics or clinical outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* a) findings on CXR that are compatible with presentations of Mycobacterium tuberculosis b) clinical symptoms, such as fever, body weight loss, night sweating, chest pain and chronic cough, that indicate active infection of pulmonary tuberculosis (TB) c) microbiological diagnosis by sputum smear and culture, bronchoalveolar lavage fluid culture, or DNA probe examination.

  d) Resolution on CXR with anti-TB regimens e) Written informed consent form prior to participation into this study

Exclusion Criteria:

* a) concurrent active disease of other chronic illnesses, such as lung cancer, chronic bronchitis and bronchial asthma b) poor physical conditions that make any examination infeasible c) participation in another trial with use of an investigated drug within on month d) use of corticosteroid or immunosuppressant drugs

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case: patients visiting the Pulmonary department of Chang Gung Memorial Hospital, Kaohsiung, Taiwan Control:healthy subjects visiting the Center of health examination at Chang Gung Memorial Hospital, Kaohsiung, Taiwan
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2006-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
susceptibility of pulmonary tuberculosis | At diagnosis

SECONDARY OUTCOMES:
clinical presentation of pulmonary TB | at diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Chih Lin, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (2):
- Taiwan (2):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung Hsien, Taiwan
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung, Taiwan